CLINICAL TRIAL: NCT04286412
Title: A SINGLE COUNTRY, MULTICENTER, OPEN-LABEL AND NON-RANDOMIZED CLINICAL TRIAL WITH NONACOG ALFA PROPHYLAXIS AND TREATMENT OF BLEEDING EPISODES IN PREVIOUSLY TREATED PATIENTS WITH MODERATELY-SEVERE TO SEVERE HEMOPHILIA B FOR A DURATION OF 8 WEEKS.
Brief Title: Nonacog Alfa Prophylaxis And Treatment Of Bleeding Episodes In Previously Treated Patients With Hemophilia B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1821059; 2020-004430-38 (EudraCT Number)
Record Dates: First submitted 2020-02-12; First posted 2020-02-27 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): At least twenty five eligible male subjects will be enrolled in the treatment arm to receive Nonacog alfa until 16 exposure days (EDs) or a period of up to 8 weeks on treatment had occurred (whichever occurs first).
  Interventions: Biological: Nonacog alfa

INTERVENTIONS:
Biological: Nonacog alfa — Nonacog alfa is indicated in India for the treatment and prophylaxis of bleeding in patients with hemophilia B (congenital factor IX deficiency).
  Other Names: BeneFIX

SUMMARY:
Nonacog alfa is indicated for the control and prevention of hemorrhagic episodes and for routine and surgical prophylaxis in patients with hemophilia B. The current single country, multi-centric, open label, non-randomized clinical trial is a post-approval study to fulfill the Central Drugs Standard Control Organization (CDSCO) request for supplementary information relating to the use of nonacog alfa in Indian subjects with hemophilia B.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥12 years to ≤65 years with a diagnosis of congenital moderately-severe to severe hemophilia B (FIX activity ≤2%).
2. Documented history of at least 50 exposure days (EDs) to FIX-containing products.
3. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative, parent(s)/legal guardian) has been informed of all pertinent aspects of the study. For minors under the age of legal consent in India, assent of the participating child needs to be documented for the age range 12 to 18 in addition to the parental informed consent.

Exclusion Criteria:

1. Prior history of inhibitor to FIX or positive inhibitor testing (≥0.6 BU/mL) during Screening. Clinical signs or symptoms of decreased response to FIX.
2. Known hypersensitivity to the active substance or any of the excipients.
3. Known allergic reaction to hamster proteins.
4. Presence of any bleeding disorder in addition to hemophilia B.
5. Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation.
6. Planned surgery within 6 months from the start of the study.
7. Unsuitable to participate in study for any other reason as assessed by the investigator; including any disorder, except for conditions associated with hemophilia B, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
8. Subjects (or a legally acceptable representative) is not able to understand study documents and study procedure.
9. Immunocompromised subjects due to human immunodeficiency virus (HIV) infection (defined as viral load above or equal to 100,000 copies/mL; and for HIV+ subjects: cluster of differentiation 4 positive (CD4+) lymphocyte count below or equal to 200/μL). HIV status and CD4+ lymphocyte count results may be obtained at screening or from available medical records; results must be not older than 6 months prior to screening.
10. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, subjects who have been previously enrolled into the study, or subjects who are Pfizer employees directly involved in the conduct of the study.
11. Planned use of any non-study medication for treatment of hemophilia (eg, other factor replacement agents, bypassing agents, or non-factor treatments [such as anti-tissue factor pathway inhibitors]).

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - K.J. Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - Sahyadri Clinical Research & Development Centre, Pune, Maharashtra
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Sahyadri Super Specialty Hospital, Pune

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1821059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in India from 10 Feb 2020 to 24 Sep 2020. A total of 25 participants were enrolled.
Pre-assignment Details: In this study, participants aged greater than or equal to 12 years to less than or equal to 65 years with congenital moderately-severe to severe hemophilia B (factor IX activity less than or equal to 2 percent) who had at least 50 exposure days (EDs) (ED was defined as a 24 hours period in which the participant was administered any FIX-containing product) to FIX-containing products were enrolled.
Groups:
- Nonacog Alfa: Participants received nonacog alfa intravenous (IV) injection as follows: Prophylactic treatment regimen: at a dose of 40 international unit per kilogram (IU/kg) (range 13 to 78 IU/kg) at intervals of 3 to 4 days in accordance with the local product document (LPD) guidelines until at least 16 exposure days or a period of up to 8 weeks on nonacog alfa treatment had occurred (whichever occurred first). For on demand (OD) treatment (infusions used to treat bleeding episodes) regimen nonacog alfa was administered at individual doses and frequency depending on the clinical effectiveness (clinical effectiveness refers to the efficacy of nonacog alfa) in individual participants as recommended in approved LPD.
Period: Overall Study
Arm/Group | Nonacog Alfa
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Groups:
- Nonacog Alfa: Participants received nonacog alfa IV injection as follows: Prophylactic treatment regimen: at a dose of 40 IU/kg (range 13 to 78 IU/kg) at intervals of 3 to 4 days in accordance with the LPD guidelines until at least 16 exposure days or a period of up to 8 weeks on nonacog alfa treatment had occurred (whichever occurred first). For OD treatment (infusions used to treat bleeding episodes) regimen nonacog alfa was administered at individual doses and frequency depending on the clinical effectiveness (clinical effectiveness refers to the efficacy of nonacog alfa) in individual participants as recommended in approved LPD.
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.44 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Factor IX (FIX) Inhibitors
Description: FIX inhibitor development was defined as an inhibitor titer >= 0.6 Bethesda units per milliliter (BU/mL) confirmed by central laboratory testing during the course of the study.
Time Frame: At Visit 4 (any 1 day between Day 52 to Day 60)
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
Percentage of participants | 0 [0.00 to 0.11]

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Medically Important Events (MIEs)
Description: An adverse events (AE) is any untoward medical occurrence in clinical investigation participant administered a product or medical device; event need not necessarily to have a causal relationship with treatment or usage. SAEs: an AE resulting in any of following outcomes/deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. MIEs: any confirmed FIX inhibitor development (titer greater than or equal to 0.6 BU/mL confirmed by central laboratory testing), thrombotic events (any event associated with the formation of a blood clot including catheter-associated thrombi and thrombotic complications) or hypersensitivity reactions (hypersensitivity reaction to a FIX product with symptoms such as hives, urticaria, tightness of chest, wheezing, hypotension, and anaphylaxis based on investigator's judgment).
Time Frame: Baseline up to 28 days after last dose of study drug (i.e, up to 116 days)
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
Participants
  SAEs | 0
  MIEs | 0

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are events between first dose of study drug and up to 116 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose of study drug (i.e, up to 116 days)
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
Participants | 3

4. Secondary Outcome: Mean Annualized Bleeding Rate (ABR)
Description: ABR: number of bleeding episodes per year. ABR for each participant = number of bleeds during treatment interval duration (TID)/(TID/365.25). Number of bleeds for each participant for ABR included all new bleeds (with unique start date and time) requiring treatment with nonacog alfa during TID. TID=date of Visit 4 (3 to 10 days after last dose) - date of Visit 2 (Day 1) +1. For participants who had Visit 4 beyond 3 (+7) days after final dose due to COVID-19 pandemic, date of final dose was used in place of date of Visit 4. For discontinued participants, date of final dose/last study visit date (whichever occurred later) was used to replace Visit 4.
Time Frame: Up to 88 Days
Population: The overall mean ABR was calculated on participants who received an on-demand infusion of Nonacog-Alfa. Since, there were no participants with bleeds, data for this outcome measure was not collected and reported.
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Annualized Total Factor Consumption (TFC) Per Participant
Description: The TFC per participant was the sum of the total amount (in international units [IU]) infused for each infusion for each participant. Annualized TFC of nonacog alfa was derived for each participant by using the following formula; Annualized TFC = (TFC / treatment interval duration)*365.25. Treatment interval duration was calculated as the number of days beginning on Visit 2 ("Day 1", provided an infusion was given) up to Visit 4 (any 1 day between Day 52 to Day 60).
Time Frame: Up to 88 Days
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Measure: Mean (Standard Deviation); unit: International units per participant
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
International units per participant | 224582.44 (75526.750)

6. Secondary Outcome: Mean Annualized Total Factor Consumption (TFC) by Weight Per Participant
Description: The total amount in international units (IU) per kilogram infused for each infusion recorded were summed to calculate the total factor consumption for each participant. Annualized TFC = (TFC / treatment interval duration)*365.25. Treatment interval duration was calculated as Date of Visit 4 - Date of Visit 2 +1. If Date of Visit 4 - Last dosing date was > 10 days then Date of Visit 4 was replaced with Last dosing date. If Date of Visit 4 was missing (due to discontinuation or any other reason), then Date of Visit 4 was replaced with last dosing date or last subject visit date, whichever was greater. International unit per kilogram= IU/kg.
Time Frame: Up to 88 days
Population: Safety analysis set included all participants who received at least 1 dose of nonacog alfa.
Measure: Mean (Standard Deviation); unit: IU/kg per participant
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 25
IU/kg per participant | 3639.27 (572.778)

7. Secondary Outcome: Mean Number of Nonacog Alfa Infusions Used to Treat Each Bleed
Description: Number of nonacog alfa infusions used to treat each bleed in participants was calculated by adding the initial (on-demand) infusion to any subsequent (on-demand) infusions for the same bleed (same bleed start date/time). On demand treatment was defined as treatment used to treat a bleeding episode.
Time Frame: Up to 88 days
Population: Since, there were no participants with bleed, therefore data for this outcome measure was not collected and analyzed.
Arm/Group | Nonacog Alfa
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (i.e, up to 116 days)
Arm/Group | Nonacog Alfa
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nonacog Alfa (N=25)
Dental caries (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT04286412/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04286412/SAP_001.pdf